CLINICAL TRIAL: NCT00783796
Title: Spirit Small Vessel Registry (SPIRIT SV)
Brief Title: SPIRIT Small Vessel Registry
Acronym: SPIRIT SV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped at 3 years. Funding for trial withdrawn by sponsor.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-383
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Results first posted 2012-01-05 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Myocardial Ischemia
Keywords: Coronary artery disease; Atherosclerosis; Myocardial ischemia
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2.25mm XIENCE V® (Experimental): Patients receiving the 2.25 mm XIENCE V® stent
  Interventions: Device: 2.25 mm XIENCE V® Everolimus Eluting Coronary Stent System

INTERVENTIONS:
Device: 2.25 mm XIENCE V® Everolimus Eluting Coronary Stent System — Treatment of a maximum of two de novo native coronary artery lesions in small vessels.

SUMMARY:
To evaluate the safety and effectiveness of the 2.25 mm XIENCE V® Everolimus Eluting Coronary Stent System (XIENCE V® EECSS) in improving coronary luminal diameter in subjects with ischemic heart disease due to a maximum of two de novo native coronary artery lesions in small vessels, each in a different epicardial vessel.

ELIGIBILITY:
General Inclusion Criteria

1. Subject must be at least 18 years of age.
2. Subject or a legally authorized representative must provide written informed consent prior to any study related procedure.
3. Subject must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or a reversible change in the electrocardiogram (ECG) consistent with ischemia).
4. Subject must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
5. Subject must agree not to participate in any other clinical study for a period of one year following the index procedure.

Angiographic Inclusion Criteria

1. One target or two (two target or one target and one non-target) de novo lesion(s), each in a different epicardial vessel.
2. If there are two target lesions or one target and one non-target lesion, both lesions must satisfy the angiographic eligibility criteria.
3. The target lesion(s) or non-target lesion must be located in a major artery or branch with a visually estimated diameter stenosis of ≥50% and < 100% with a TIMI flow of ≥1.
4. The target lesion(s) or non-target lesion must be located in a native coronary artery with a reference vessel diameter by visual estimation of: Target Lesion: ≥ 2.25 mm to < 2.5 mm for treatment by the 2.25 mm XIENCE V® EECS.

   Non-target Lesion: ≥2.5 mm to ≤4.25 mm for treatment by the commercial XIENCE V® EECS.
5. The target lesion(s) or non-target lesion must be located in a native coronary artery with a lesion length by visual estimation of ≤28 mm.

General Exclusion Criteria

1. Subject has had a known diagnosis of acute myocardial infarction (AMI) preceding the index procedure (CK-MB (creatine kinase myocardial-band isoenzyme) ≥2 times the upper limit of normal) and CK and CK-MB levels have not returned to within normal limits at the time of procedure.
2. The subject is currently experiencing clinical symptoms consistent with new onset AMI, such as nitrate-unresponsive prolonged chest pain with ischemic ECG changes.
3. Subject has current unstable cardiac arrhythmias associated with hemodynamic instability.
4. Subject has a known left ventricular ejection fraction (LVEF) < 30% (LVEF may be obtained at the time of the index procedure if the value is unknown and if necessary).
5. Subject has received coronary brachytherapy in any epicardial vessel.
6. Subject has received any organ transplant or is on a waiting list for any organ transplant.
7. Subject is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or within one year after the index procedure.
8. Subject is receiving or scheduled to receive planned radiation therapy to the chest or mediastinum.
9. Subject is receiving immunosuppressant therapy or has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus etc.).
10. Subject is receiving chronic anticoagulation therapy (e.g., heparin, coumadin).
11. Subjects who will require Low Molecular Weight Heparin (LMWH) post-procedure.
12. Subject has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/ticlopidine, everolimus, cobalt, chromium, nickel, tungsten, acrylic and fluoropolymers or contrast sensitivity that cannot be adequately pre-medicated.
13. Elective surgery is planned within 12 months after the procedure that will require discontinuing either aspirin or clopidogrel.
14. Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC (white blood cell) of < 3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis).
15. Subject has known renal insufficiency (eg, serum creatinine level ≥ 2.5 mg/dL, or on dialysis).
16. Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
17. Subject has had a cerebrovascular accident/stroke or transient ischemic neurological attack (TIA) within the past six months.
18. Subject has had a significant gastro-intestinal or significant urinary bleed within the past six months.
19. Subject has extensive peripheral vascular disease that precludes safe 6 French sheath insertion.
20. Subject has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year).
21. Subject is currently participating in another clinical study that has not yet completed its primary endpoint.
22. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.

Angiographic Exclusion Criteria

1. Target lesion(s) or non-target lesion located within an arterial or saphenous vein graft or distal to a diseased (vessel irregularity per angiogram and > 20% stenosed lesion by visual estimation) arterial or saphenous vein graft.
2. Target lesion(s) or non-target lesion involving a bifurcation with a side branch ≥2 mm in diameter and/or ostial lesion > 40% stenosed by visual estimation or side branch requiring protection guide wire, or side branch requiring dilatation.
3. Total occlusion (TIMI flow 0), prior to crossing with the wire.
4. Another lesion requiring revascularization is located in the same epicardial vessel of either the target or non-target lesion.
5. Restenotic lesion.
6. Aorto-ostial lesion (within 3 mm of the aorta junction).
7. Left main location.
8. Lesion located within 2 mm of the origin of the LAD (left anterior descending) or LCX (left coronary artery)
9. Extreme angulation (≥90°) or excessive tortuosity (≥ two 45° angles) proximal to or within the target or non-target lesion.
10. Heavy calcification proximal to or within the target or non-target lesion(s).
11. Target or non-target vessel contains thrombus as indicated in the angiographic images.
12. Target lesion(s) or non-target lesion have a high probability that a procedure other than pre-dilatation and stenting will be required at the time of index procedure for treating the target and non-target vessel(s) (e.g. atherectomy, cutting balloon).
13. Target or non-target vessel(s) have previously been treated with percutaneous intervention (e.g. balloon angioplasty, stent, cutting balloon, atherectomy) < 9 months prior to index procedure.
14. A vessel not intended to be treated with a 2.25 mm XIENCE V® EECS or commercial sizes of XIENCE V® EECS that was previously treated with any type of PCI (percutaneous coronary intervention) < 90 days prior to the index procedure.
15. Additional clinically significant lesion(s) (e.g., %DS (diameter stenosis) ≥ 50%) is present in any vessel or side branch for which PCI may be required < 90 days after the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco A. Costa, MD, PhD, Principal Investigator — Case Western University Hospital, Cleveland, OH
Locations (34):
- United States (34):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - St. Anthony Hospital, Rockford, Illinois
  - St. John's Hospital / Prairie Education & Research Cooperative, Springfield, Illinois
  - Union Memorial Hospital, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - St. Joseph Medical Center, Towson, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Joseph Mercy Hospital, Ypsilanti, Michigan
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - St. Patrick Hospital, Missoula, Montana
  - Cooper Health System, Camden, New Jersey
  - Gotham Cardiovascular Reasearch, PC. (St. Vincent's Medical Center-closing, pts moved), New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - WakeMed Hospital, Raleigh, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - EMH Regional Medical Center, Elyria, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Baptist West Hospital, Knoxville, Tennessee
  - Northwest Texas Healthcare System, Amarillo, Texas
  - Mother Frances Hospital, Tyler, Texas
  - Overlake Hospital Medical Center, Bellevue, Washington
  - St. Joseph Hospital, Bellingham, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 150 subjects were recruited at 33 sites from the general interventional cardiology population. Dates of recruitment: 12/08/08 through 11/04/09.
Pre-assignment Details: Subjects were screened for study eligibility by a member of the study team. Subjects meeting eligibility criteria were asked to sign an informed consent form. Pre-procedure angiography was used for final assessment of eligibility.
Groups:
- 2.25mm XIENCE V®: Patients receiving the 2.25 mm XIENCE V® Everolimus Eluting Coronary Stent System (EECSS)
Period: Overall Study
Arm/Group | 2.25mm XIENCE V®
Started | 150
Completed | 144
Not Completed | 6
Not completed — Did not receive any stent | 4
Not completed — Received non-XIENCE V stent | 1
Not completed — Received commercial XIENCE V stent | 1

BASELINE CHARACTERISTICS:
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 85
  >=65 years | 65
Age, Continuous [Mean (Standard Deviation); unit: years] — This calculation is based on the FAS population (144 subjects), this removes 6 subjects who did not receive the 2.25mm XIENCE V® stent.
  years | 62.97 (10.59)
Sex/Gender, Customized [Number; unit: participants] — One participant was de-registered from the study without recording their gender. The total number of participants is 150, however there is only gender data for 149 subjects
  participants
    Female | 57
    Male | 92
Region of Enrollment [Number; unit: participants]
  United States | 150

OUTCOME MEASURES:

1. Primary Outcome: Composite Rate of Cardiac Death, Target Vessel Myocardial Infarction (MI) (Per Protocol Definition) & Clinically Indicated Target Lesion Revascularization (CI-TLR).
Description: This endpoint is a composite of cardiac death, target vessel myocardial infarction per protocol definition, and clinically-indicated target lesion revascularization.
Time Frame: 1 year
Population: The number of participants analyzed is based on FAS population, defined as subjects who have received the investigational study device (2.25 mm XIENCE V stent) and excludes subjects who are truly lost-to-follow-up, defined as subjects who are lost to follow-up through given timepoint without any DMR event (all death, all MI, all revascularization).
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 136
Percentage of Participants | 8.1

2. Primary Outcome: Composite Rate of Cardiac Death, Target Vessel Myocardial Infarction (MI) (Per Protocol Definition) & Clinically Indicated Target Lesion Revascularization (CI-TLR).
Description: as for outcome 1
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 132
Percentage of Participants | 8.3

3. Primary Outcome: Composite Rate of Cardiac Death, Target Vessel Myocardial Infarction (MI) (Per Protocol Definition) & Clinically Indicated Target Lesion Revascularization (CI-TLR).
Description: as for outcome 1
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 132
Percentage of Participants | 12.1

4. Secondary Outcome: Device Success (Per Lesion Basis, for Target Lesions Treated by 2.25 mm XIENCE V EECS With or Without Planned Overlap)
Description: Successful delivery and deployment of the first study stent intended to be implanted at the intended target lesion (or intended first and second investigational stents for overlapping stents), successful withdrawal of the stent delivery system, and attainment of final residual stenosis of <50%.
Time Frame: From start of index procedure to end of index procedure
Population: Based on Intent To Treat (ITT) population, defined as subjects enrolled in the study, regardless of the treatment actually received, and excluding de-registered subjects
Measure: Number; unit: Percentage of Lesions
Units Other Than Participants: Lesions
Groups:
- 2.25mm XIENCE V®: Based on Intent To Treat (ITT) population, defined as subjects enrolled in the study, regardless of the treatment actually received, and excluding de-registered subjects
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 146
Number analyzed (Lesions) | 149
Percentage of Lesions | 95.21

5. Secondary Outcome: Procedural Success (Per Subject Basis, for ALL Target and Non-target Lesions)
Description: Achievement of a final in-stent diameter stenosis of <50% using the study device, without the occurence of cardiac death, target vessel myocardial infarction per protocol definition, or repeat revascularization of the target lesion during the hospital stay up to 7 days.
Time Frame: From the start of index procedure to end of index procedure
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 145
Percentage of Participants | 97.93

6. Secondary Outcome: In-Stent Late Loss
Description: In-stent minimum lumen diameter (MLD) post-procedure minus in-stent MLD at angiographic follow-up.
Time Frame: 240 days
Population: Based on Angiographic Cohort Full Analysis Set (FAS) population, defined as subjects in the Angiographic Cohort who have received the investigational study device (2.25 mm XIENCE V stent).
Measure: Mean (Standard Deviation); unit: Millimeters
Groups:
- 2.25mm XIENCE V®: Patients in the Angiographic Cohort receiving the 2.25 mm XIENCE V Stent
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 52
Millimeters | 0.20 (0.40)

7. Secondary Outcome: In-segment Late Loss (LL)
Description: In-segment minimum lumen diameter (MLD) post-procedure minus in-segment MLD at angiographic follow-up.
Time Frame: 240 Days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 52
Millimeters | 0.16 (0.41)

8. Secondary Outcome: Proximal Late Loss
Description: Proximal minimum lumen diameter (MLD) post-procedure minus proximal MLD at angiographic follow-up (proximal defined as 5 mm of healthy tissue proximal to stent placement).
Time Frame: 240 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 34
Millimeter | 0.21 (0.35)

9. Secondary Outcome: Distal Late Loss
Description: Distal minimum lumen diameter (MLD) post-procedure minus distal MLD at angiographic follow-up (distal defined as 5 mm of healthy tissue distal to stent placement).
Time Frame: 240 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 45
Millimeter | 0.00 (0.28)

10. Secondary Outcome: In-stent % Diameter Stenosis
Description: Value calculated as 100*(1-MLD/RVD) where MLD is in-stent minimum lumen diameter and RVD is in-stent reference vessel diameter.
Time Frame: 240 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 52
Percentage | 12.86 (19.58)

11. Secondary Outcome: In-segment % Diameter Stenosis
Description: Value calculated as 100*(1-MLD/RVD) where MLD is in-segment minimum lumen diameter and RVD is in-segment reference vessel diameter.
Time Frame: 240 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 52
Percentage | 20.85 (22.53)

12. Secondary Outcome: Proximal % Diameter Stenosis
Description: Value calculated as 100*(1-MLD/RVD) where MLD is minimum lumen diameter and RVD is reference vessel diameter in 5 mm of healthy tissue proximal to stent placement.
Time Frame: 240 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 37
Percentage | 14.31 (13.16)

13. Secondary Outcome: Distal % Diameter Stenosis
Description: Value calculated as 100*(1-MLD/RVD) where MLD is minimum lumen diameter and RVD is reference vessel diameter in 5 mm of healthy tissue distal to stent placement.
Time Frame: 240 days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 46
Percentage | 10.4 (8.45)

14. Secondary Outcome: In-stent Angiographic Binary Restenosis (ABR) Rate
Description: Percentage of patients with target lesions with ≥ 50% in-stent % diameter stenosis at angiographic follow-up.
Time Frame: 240 days
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 52
Percentage of Participants | 3.8 [0.47 to 13.21]

15. Secondary Outcome: In-segment Angiographic Binary Restenosis (ABR) Rate
Description: Percentage of patients with target lesions with ≥ 50% in-segment % diameter stenosis at angiographic follow-up.
Time Frame: 240 days
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 52
Percentage of Participants | 9.6 [3.20 to 21.03]

16. Secondary Outcome: Proximal Angiographic Binary Restenosis (ABR) Rate
Description: Percentage of patients with target lesions with ≥ 50% diameter stenosis in 5 mm of healthy tissue proximal to stent placement at angiographic follow-up.
Time Frame: 240 days
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 37
Percentage of Participants | 2.7 [0.07 to 14.16]

17. Secondary Outcome: Distal Angiographic Binary Restenosis (ABR) Rate
Description: Percentage of patients with target lesions with ≥ 50% diameter stenosis in 5 mm of healthy tissue distal to stent placement at angiographic follow-up.
Time Frame: 240 days
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 46
Percentage of Participants | 0.0 [0.00 to 7.71]

18. Secondary Outcome: All Death (Cardiac, Vascular, Non-cardiovascular)
Description: All death, including death from cardiac, vascular, and non-cardiovascular causes.
Time Frame: 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 144
Percentage of Participants | 0.7 [0.02 to 3.81]

19. Secondary Outcome: All Death (Cardiac, Vascular, Non-cardiovascular)
Description: All death, including death from cardiac, vascular, and non-cardiovascular causes.
Time Frame: 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 139
Percentage of Participants | 1.4 [0.17 to 5.10]

20. Secondary Outcome: All Death (Cardiac, Vascular, Non-cardiovascular)
Description: All death, including death from cardiac, vascular, and non-cardiovascular causes.
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 136
Percentage of Participants | 1.5 [0.18 to 5.21]

21. Secondary Outcome: All Death (Cardiac, Vascular, Non-cardiovascular)
Description: All death, including death from cardiac, vascular, and non-cardiovascular causes.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 133
percentage of participants | 1.5 [0.18 to 5.33]

22. Secondary Outcome: All Death (Cardiac, Vascular, Non-cardiovascular)
Description: All death, including death from cardiac, vascular, and non-cardiovascular causes (per protocol).
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 132
percentage of participants | 3.8 [1.24 to 8.62]

23. Secondary Outcome: Target Vessel MI - Q-wave and Non Q-wave (Per Protocol)
Description: Target vessel myocardial infarction (MI) (MI not clearly attributable to a non-target vessel), including Q-wave MI (new pathologic Q waves) and Non Q-wave MI (elevation of CK to ≥ two times the upper limit normal with elevated CK-MB in the absence of new pathological Q waves).
Time Frame: 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 144
Percentage of Participants | 1.4 [0.17 to 4.93]

24. Secondary Outcome: Target Vessel MI - Q-wave and Non Q-wave (Per Protocol)
Description: as for outcome 23
Time Frame: 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 139
Percentage of Participants | 1.4 [0.17 to 5.10]

25. Secondary Outcome: Target Vessel MI - Q-wave and Non Q-wave (Per Protocol)
Description: as for outcome 23
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 136
Percentage of Participants | 1.5 [0.18 to 5.21]

26. Secondary Outcome: Target Vessel MI - Q-wave and Non Q-wave (Per Protocol)
Description: as for outcome 23
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 133
percentage of participants | 1.5 [0.18 to 5.33]

27. Secondary Outcome: Target Vessel MI - Q-wave and Non Q-wave (Per Protocol)
Description: as for outcome 23
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 132
percentage of participants | 1.5 [0.18 to 5.37]

28. Secondary Outcome: Stent Thrombosis (ARC Defined)
Description: ARC defined: Stent Thrombosis as per Academic Research Consortium standardized definitions (Circulation 2007;115:2344-2351). Result includes Definite/Probable/Possible.
Time Frame: 0 to 1 day (Acute)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 142
Percentage of Participants | 0.0

29. Secondary Outcome: Stent Thrombosis (ARC Defined)
Description: as for outcome 28
Time Frame: greater than 1 day to 30 days (Subacute)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 140
Percentage of Participants | 0.7

30. Secondary Outcome: Stent Thrombosis (ARC Defined)
Description: Stent Thrombosis as per Academic Research Consortium standardized definitions (Circulation 2007;115:2344-2351). Result includes Definite/Probable/Possible.
Time Frame: 31 days - 393 days (Late)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 135
Percentage of Participants | 1.5

31. Secondary Outcome: Stent Thrombosis (ARC Defined)
Description: as for outcome 30
Time Frame: >1 year (Very late)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 130
Percentage of Participants | 0.0

32. Secondary Outcome: Stent Thrombosis (ARC Defined)
Description: as for outcome 30
Time Frame: 394 - 758 days (Very Late)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 129
Percentage of Participants | 0.0

33. Secondary Outcome: Stent Thrombosis (ARC Defined)
Description: as for outcome 30
Time Frame: 394 - 1123 days (Very Late)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 128
Percentage of Participants | 0.78

34. Secondary Outcome: Stent Thrombosis (ARC Defined)
Description: as for outcome 30
Time Frame: Overall (0 - 393 days)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 138
Percentage of Participants | 2.17

35. Secondary Outcome: Stent Thrombosis (ARC Defined)
Description: as for outcome 30
Time Frame: Overall (0 - 758 days)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 131
Percentage of Participants | 2.29

36. Secondary Outcome: Stent Thrombosis (ARC Defined)
Description: as for outcome 30
Time Frame: Overall (0 - 1123 days)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 130
Percentage of Participants | 3.08

37. Secondary Outcome: Stent Thrombosis (Protocol Defined)
Description: Stent Thrombosis per protocol categorized as acute (≤1 day), subacute (>1 day and ≤30 days), and late (>30 days), and defined as clinical presentation of acute coronary syndrome with angiographic evidence of stent thrombosis, or in absence of angiography, any unexplained death at any time or acute myocardial infarction* (ST segment elevation or new Q-wave) in the distribution of the target lesion within 30 days of the index procedure. (*Non-specific ST/T changes and cardiac enzymes do not suffice.). Result includes Definite/Probable/Possible.
Time Frame: 0 to 1 day (Acute)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 142
Percentage of Participants | 0.0

38. Secondary Outcome: Stent Thrombosis (Protocol Defined)
Description: as for outcome 37
Time Frame: > 1 day to 30 days (Subacute)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 140
Percentage of Participants | 0.7

39. Secondary Outcome: Stent Thrombosis (Protocol Defined)
Description: as for outcome 37
Time Frame: 31 days to 393 days (Late)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 135
Percentage of Participants | 1.5

40. Secondary Outcome: Stent Thrombosis (Protocol Defined)
Description: as for outcome 37
Time Frame: 31 - 758 days (Late)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 130
Percentage of Participants | 1.5

41. Secondary Outcome: Stent Thrombosis (Protocol Defined)
Description: as for outcome 37
Time Frame: 31 - 1123 days (Late)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 129
Percentage of Participants | 2.3

42. Secondary Outcome: Stent Thrombosis (Protocol Defined)
Description: as for outcome 37
Time Frame: Overall (0 - 393 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 138
percentage of participants | 2.2

43. Secondary Outcome: Stent Thrombosis (Protocol Defined)
Description: as for outcome 37
Time Frame: Overall (0 - 758 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 132
percentage of participants | 2.27

44. Secondary Outcome: Stent Thrombosis (Protocol Defined)
Description: as for outcome 37
Time Frame: Overall (0 - 1123 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 130
percentage of participants | 3.1

45. Secondary Outcome: All Death/ All MI/All Coronary Revascularization
Description: This endpoint is a composite of all death, all myocardial infarction per protocol definition, and all revascularization.
Time Frame: 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 144
Percentage of Participants | 3.5 [1.14 to 7.92]

46. Secondary Outcome: All Death/ All MI/All Coronary Revascularization
Description: This endpoint is a composite of all death, all myocardial infarction per protocol definition, and all revascularization.
Time Frame: 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 139
Percentage of Participants | 15.1 [9.60 to 22.16]

47. Secondary Outcome: All Death/ All MI/All Coronary Revascularization
Description: This endpoint is a composite of all death, all myocardial infarction per protocol definition, and all revascularization.
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 136
Percentage of Participants | 16.9 [11.03 to 24.29]

48. Secondary Outcome: All Death/ All MI/All Coronary Revascularization
Description: This endpoint is a composite of all death, all myocardial infarction per protocol definition, and all revascularization.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 133
percentage of participants | 22.6 [15.77 to 30.61]

49. Secondary Outcome: All Death/ All MI/All Coronary Revascularization
Description: This endpoint is a composite of all death, all myocardial infarction per protocol definition, and all revascularization.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 132
percentage of participants | 26.5 [19.21 to 34.9]

50. Secondary Outcome: Cardiac Death/ All MI /CI-TLR
Description: This endpoint is a composite of cardiac death, all myocardial infarction (MI)per protocol definition, and clinically-indicated target lesion revascularization (CI-TLR).
Time Frame: 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 144
Percentage of Participants | 2.1 [0.43 to 5.97]

51. Secondary Outcome: Cardiac Death/ All MI /CI-TLR
Description: as for outcome 50
Time Frame: 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 139
Percentage of Participants | 7.2 [3.5 to 12.83]

52. Secondary Outcome: Cardiac Death/ All MI /CI-TLR
Description: as for outcome 50
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 136
Percentage of Participants | 8.1 [4.11 to 14.01]

53. Secondary Outcome: Cardiac Death/ All MI /CI-TLR
Description: as for outcome 50
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 133
percentage of participants | 8.3 [4.2 to 14.32]

54. Secondary Outcome: Cardiac Death/ All MI /CI-TLR
Description: as for outcome 50
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 132
percentage of participants | 12.1 [7.09 to 18.94]

55. Secondary Outcome: Cardiac Death/MI
Description: This endpoint is a composite of cardiac death and all myocardial infarction per protocol definition.
Time Frame: 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 144
Percentage of Participants | 2.1 [0.43 to 5.97]

56. Secondary Outcome: Cardiac Death/MI
Description: This endpoint is a composite of cardiac death and all myocardial infarction per protocol definition.
Time Frame: 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 139
Percentage of Participants | 2.9 [0.79 to 7.20]

57. Secondary Outcome: Cardiac Death/MI
Description: This endpoint is a composite of cardiac death and all myocardial infarction per protocol definition.
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 136
Percentage of Participants | 2.9 [0.81 to 7.36]

58. Secondary Outcome: Cardiac Death/MI
Description: This endpoint is a composite of cardiac death and all myocardial infarction per protocol definition.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 133
percentage of participants | 3.0 [0.83 to 7.52]

59. Secondary Outcome: Cardiac Death/MI
Description: This endpoint is a composite of cardiac death and all myocardial infarction per protocol definition.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 132
percentage of participants | 5.3 [2.16 to 10.62]

60. Secondary Outcome: All Coronary Revascularization (TVR and Non-TVR)
Description: Includes any revascularization intervention after the index procedure by any means (percutaneous or bypass surgery), including intervention to the target vessel, and intervention to a vessel other than the target vessel.
Time Frame: 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 144
Percentage of Participants | 2.1 [0.43 to 5.97]

61. Secondary Outcome: All Coronary Revascularization (TVR and Non-TVR)
Description: as for outcome 60
Time Frame: 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 139
Percentage of Participants | 12.9 [7.86 to 19.69]

62. Secondary Outcome: All Coronary Revascularization (TVR and Non-TVR)
Description: as for outcome 60
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 136
Percentage of Participants | 14.7 [9.22 to 21.79]

63. Secondary Outcome: All Coronary Revascularization (TVR and Non-TVR)
Description: as for outcome 60
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 133
percentage of participants | 20.3 [13.83 to 28.14]

64. Secondary Outcome: All Coronary Revascularization (TVR and Non-TVR)
Description: Includes any revascularization intervention after the index procedure by any means (percutaneous or bypass surgery), including intervention to the target vessel, and intervention to a vessel other than the target vessel (per protocol).
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 132
percentage of participants | 23.5 [16.55 to 31.65]

65. Secondary Outcome: All TVR (CI and Non-CI)
Description: Includes any repeat revascularization intervention after the index procedure by any means (percutaneous or bypass surgery) in the target vessel from the index procedure.
Time Frame: 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 144
Percentage of Participants | 1.4 [0.17 to 4.93]

66. Secondary Outcome: All TVR (CI and Non-CI)
Description: as for outcome 65
Time Frame: 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 139
Percentage of Participants | 8.6 [4.54 to 14.59]

67. Secondary Outcome: All TVR (CI and Non-CI)
Description: as for outcome 65
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 136
Percentage of Participants | 10.3 [5.74 to 16.67]

68. Secondary Outcome: All TVR (CI and Non-CI)
Description: as for outcome 65
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 133
percentage of participants | 11.3 [6.45 to 17.92]

69. Secondary Outcome: All TVR (CI and Non-CI)
Description: Includes any repeat revascularization intervention after the index procedure by any means (percutaneous or bypass surgery) in the target vessel from the index procedure (per protocol).
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 132
percentage of participants | 13.6 [8.29 to 20.69]

70. Secondary Outcome: All TLR (CI and Non-CI)
Description: Includes any repeat revascularization intervention after the index procedure by any means (percutaneous or bypass surgery) of the target lesion from the index procedure. This includes interventions classified as clinically indicated, and also includes interventions classified as not clinically indicated.
Time Frame: 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 144
Percentage of Participants | 0.7 [0.02 to 3.81]

71. Secondary Outcome: All TLR (CI and Non-CI)
Description: as for outcome 70
Time Frame: 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 139
Percentage of Participants | 5.8 [2.52 to 11.03]

72. Secondary Outcome: All TLR (CI and Non-CI)
Description: as for outcome 70
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 136
Percentage of Participants | 6.6 [3.07 to 12.19]

73. Secondary Outcome: All TLR (CI and Non-CI)
Description: as for outcome 70
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 133
percentage of participants | 6.8 [3.14 to 12.46]

74. Secondary Outcome: All TLR (CI and Non-CI)
Description: Includes any repeat revascularization intervention after the index procedure by any means (percutaneous or bypass surgery) of the target lesion from the index procedure. This includes interventions classified as clinically indicated, and also includes interventions classified as not clinically indicated (per protocol).
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 132
percentage of participants | 8.3 [4.23 to 14.42]

75. Secondary Outcome: Clinically Indicated Target Vessel Revascularization (TVR)
Description: Includes clinically indicated repeat revascularization after the index procedure by any means (percutaneous or bypass surgery), of the target vessel. Classification as clinically indicated is done prospectively and verified by angiographic core lab measurement, and requires ≥50% diameter stenosis with ischemic signs or symptoms (positive history of angina pectoris or objective signs of ischemia at rest (ECG changes) or during exercise test or abnormal invasive cardiac functional diagnostic test), or ≥70% diameter stenosis in the absence of the above-mentioned ischemic signs or symptoms.
Time Frame: 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 144
Percentage of Participants | 1.4 [0.17 to 4.93]

76. Secondary Outcome: Clinically Indicated Target Vessel Revascularization
Description: as for outcome 75
Time Frame: 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 139
Percentage of Participants | 7.2 [3.50 to 12.83]

77. Secondary Outcome: Clinically Indicated Target Vessel Revascularization
Description: as for outcome 75
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 136
Percentage of Participants | 8.8 [4.64 to 14.91]

78. Secondary Outcome: Clinically Indicated Target Vessel Revascularization
Description: as for outcome 75
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 133
percentage of participants | 9.8 [5.31 to 16.13]

79. Secondary Outcome: Clinically Indicated Target Vessel Revascularization
Description: Includes clinically indicated repeat revascularization after the index procedure by any means (percutaneous or bypass surgery), of the target vessel. Classification as clinically indicated is done prospectively and verified by angiographic core lab measurement, and requires ≥50% diameter stenosis with ischemic signs or symptoms (positive history of angina pectoris or objective signs of ischemia at rest (ECG changes) or during exercise test or abnormal invasive cardiac functional diagnostic test), or ≥70% diameter stenosis in the absence of the above-mentioned ischemic signs or symptoms (per protocol).
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 132
percentage of participants | 12.1 [7.09 to 18.94]

80. Secondary Outcome: Clinically Indicated Target Lesion Revascularization (CI-TLR)
Description: Includes clinically indicated repeat revascularization after the index procedure by any means (percutaneous or bypass surgery) of the target lesion. Classification as clinically indicated is done prospectively and verified by angiographic core lab measurement, and requires ≥50% diameter stenosis with ischemic signs or symptoms (positive history of angina pectoris or objective signs of ischemia at rest (ECG changes) or during exercise test or abnormal invasive cardiac functional diagnostic test), or ≥70% diameter stenosis in the absence of the above-mentioned ischemic signs or symptoms.
Time Frame: 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 144
Percentage of Participants | 0.0 [0.0 to 2.53]

81. Secondary Outcome: Clinically Indicated Target Lesion Revascularization (CI-TLR)
Description: as for outcome 80
Time Frame: 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 139
Percentage of Participants | 4.3 [1.60 to 9.16]

82. Secondary Outcome: Clinically Indicated Target Lesion Revascularization (CI-TLR)
Description: as for outcome 80
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 136
Percentage of Participants | 5.1 [2.09 to 10.32]

83. Secondary Outcome: Clinically Indicated Target Lesion Revascularization (CI-TLR)
Description: as for outcome 80
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 133
percentage of participants | 5.3 [2.14 to 10.54]

84. Secondary Outcome: Clinically Indicated Target Lesion Revascularization (CI-TLR)
Description: Includes clinically indicated repeat revascularization after the index procedure by any means (percutaneous or bypass surgery) of the target lesion. Classification as clinically indicated is done prospectively and verified by angiographic core lab measurement, and requires ≥50% diameter stenosis with ischemic signs or symptoms (positive history of angina pectoris or objective signs of ischemia at rest (ECG changes) or during exercise test or abnormal invasive cardiac functional diagnostic test), or ≥70% diameter stenosis in the absence of the above-mentioned ischemic signs or symptoms (per protocol).
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 132
percentage of participants | 6.8 [3.16 to 12.55]

85. Secondary Outcome: Non Target Vessel MI (Q-wave, Non Q-wave)(Per Protocol)
Description: Non target vessel myocardial infarction (MI) (MI clearly attributable to a non-target vessel), including Q-wave MI (new pathologic Q waves) and Non Q-wave MI (elevation of CK to ≥ two times the upper limit normal with elevated CK-MB in the absence of new pathological Q waves).
Time Frame: 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 144
Percentage of Participants | 0.0 [0.0 to 2.53]

86. Secondary Outcome: Non Target Vessel MI (Q-wave, Non Q-wave)(Per Protocol)
Description: as for outcome 85
Time Frame: 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 139
Percentage of Participants | 0.0 [0.0 to 2.62]

87. Secondary Outcome: Non Target Vessel MI (Q-wave, Non Q-wave)(Per Protocol)
Description: as for outcome 85
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 136
Percentage of Participants | 0.0 [0.0 to 2.68]

88. Secondary Outcome: Non Target Vessel MI (Q-wave, Non Q-wave)(Per Protocol)
Description: as for outcome 85
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 133
percentage of participants | 0.0 [0.0 to 2.74]

89. Secondary Outcome: Non Target Vessel MI (Q-wave, Non Q-wave)(Per Protocol)
Description: as for outcome 85
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 132
percentage of participants | 0.0 [0.00 to 2.76]

90. Secondary Outcome: Target Vessel MI - Q-wave and Non Q-wave (Per ARC)
Description: ARC defined target vessel MI (MI not clearly attributable to a non-target vessel): Myocardial Infarction as per Academic Research Consortium standardized definitions (Circulation 2007;115:2344- 2351).
Time Frame: 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 144
Percentage of Participants | 6.3 [2.90 to 11.53]

91. Secondary Outcome: Target Vessel MI - Q-wave and Non Q-wave (Per ARC)
Description: as for outcome 90
Time Frame: 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 139
Percentage of Participants | 6.5 [3.0 to 11.94]

92. Secondary Outcome: Target Vessel MI - Q-wave and Non Q-wave (Per ARC)
Description: as for outcome 90
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 136
Percentage of Participants | 6.6 [3.07 to 12.19]

93. Secondary Outcome: Target Vessel MI - Q-wave and Non Q-wave (Per ARC)
Description: as for outcome 90
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 134
percentage of participants | 6.7 [3.12 to 12.37]

94. Secondary Outcome: Target Vessel MI - Q-wave and Non Q-wave (Per ARC)
Description: as for outcome 90
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 133
percentage of participants | 7.5 [3.66 to 13.39]

95. Secondary Outcome: Non Target Vessel MI- Q-wave, Non Q-wave (Per ARC)
Description: ARC defined non-target vessel MI (MI clearly attributable to a non-target vessel): Myocardial Infarction as per Academic Research Consortium standardized definitions (Circulation 2007;115:2344- 2351).
Time Frame: 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 144
Percentage of participants | 0.0 [0.0 to 2.53]

96. Secondary Outcome: Non Target Vessel MI- Q-wave, Non Q-wave (Per ARC)
Description: as for outcome 95
Time Frame: 240 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 139
Percentage of participants | 1.4 [0.17 to 5.10]

97. Secondary Outcome: Non Target Vessel MI- Q-wave, Non Q-wave (Per ARC)
Description: as for outcome 95
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 136
Percentage of participants | 1.5 [0.18 to 5.21]

98. Secondary Outcome: Non Target Vessel MI- Q-wave, Non Q-wave (Per ARC)
Description: as for outcome 95
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 134
percentage of participants | 1.5 [0.18 to 5.29]

99. Secondary Outcome: Non Target Vessel MI- Q-wave, Non Q-wave (Per ARC)
Description: as for outcome 95
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2.25mm XIENCE V®
Number analyzed (Participants) | 133
percentage of participants | 4.5 [1.67 to 9.56]

ADVERSE EVENTS:
Time Frame: 0 to 1123 Day Serious Site-Reported, Un-Adjudicated Adverse Events Regardless of Relationship to the Device.
Description: The number of participants at risk does not always remain at 144 through the 3 years because 5 participants terminated sometime between 0-1123 days without any event and had no further information. These 5 patients were excluded from the denominator (this is a conservative approach) and at no time were event subjects excluded from the calculation.
Arm/Group | 2.25mm XIENCE V®
Serious Adverse Events (participants affected / at risk) | 79/139
Other Adverse Events (participants affected / at risk) | 83/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.25mm XIENCE V® (N=139)
Deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 5 (5)
Angina pectoris (Cardiac disorders) | 27 (33)
Angina unstable (Cardiac disorders) | 8 (8)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 6 (8)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 4 (5)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 6 (7)
Coronary artery dissection (Cardiac disorders) | 1 (1)
Coronary artery perforation (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 6 (6)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1)
Blindness (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Catheter site haematoma (General disorders) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 6 (11)
Sarcoidosis (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Pyelonephritis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Wound infection staphylococcal (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 5 (6)
Mechanical complication of implant (Injury, poisoning and procedural complications) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1)
Cardiac enzymes increased (Investigations) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Convulsion (Nervous system disorders) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 2 (2)
Post-traumatic headache (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 2 (3)
Syncope (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 4 (4)
Vertigo (Nervous system disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (2)
Calculus bladder (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Carotid arteriosclerosis (Vascular disorders) | 1 (1)
Carotid artery disease (Vascular disorders) | 2 (2)
Carotid artery occlusion (Vascular disorders) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 2 (3)
Gastric ulcer haemorrhage (Vascular disorders) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1)
Intestinal haemorrhage (Vascular disorders) | 1 (1)
Renal artery stenosis (Vascular disorders) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.25mm XIENCE V® (N=139)
Angina pectoris (Cardiac disorders) | 39 (50)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7)
Fatigue (General disorders) | 9 (10)
Non-cardiac chest pain (General disorders) | 25 (30)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8)
Dizziness (Nervous system disorders) | 13 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (16)
Contusion (Vascular disorders) | 7 (8)
Hypertension (Vascular disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days